CLINICAL TRIAL: NCT01967095
Title: A Phase 1 Trial of Low Dose Daily Erlotinib in Combination With High Dose Twice Weekly Erlotinib in Patients With EGFR-Mutant Lung Cancer
Brief Title: Low Dose Daily Erlotinib in Combination With High Dose Twice Weekly Erlotinib in Patients With EGFR-Mutant Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Astellas Pharma US, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-278
Record Dates: First submitted 2013-10-15; First posted 2013-10-22 (Estimated); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: EGFR-Mutant Lung Cancer
Keywords: Erlotinib; 12-278; CNS involvement
MeSH Terms: interventions — Erlotinib Hydrochloride; Lead

ARMS (1):
- erlotinib (Experimental): This protocol is a phase 1, single arm, open label study of combination daily low dose erlotinib plus twice weekly high dose erlotinib in patients with EGFR-Mutant lung cancer who have not yet received erlotinib or gefitinib. Six dose levels are planned for escalation, with the pulse dose erlotinib increasing.
  Expansion cohort A: Treat an additional 19 pts at the MTD with CNS involvement at diagnosis
  Interventions: Drug: erlotinib

INTERVENTIONS:
Drug: erlotinib — Cycle 1, week 1 (D1-D7) will consist of pulse dose erlotinib on D1 & D2 without daily low dose erlotinib on D3-7. For all subsequent weeks, patients will take high dose erlotinib on D1 & D2, & will receive erlotinib 50 mg oral daily x 5 days on days 3-7. On days 1 & 2, patients will take one of the following doses of erlotinib, depending on the dose cohort they are enrolled in: Dose level 1 600 mg oral daily on D1, D2 Dose level 2 750 mg oral daily on D1, D2 Dose level 3 900 mg oral daily on D1, D2 Dose level 4 1050 mg oral daily on D1, D2. An additional Dose -1 (pulse dose erlotinib on D1, D2 with 25 mg oral daily x 5 days in D3-D7) will be reserved, in the unlikely situation that Dose 1 is proved too toxic. If Dose -1 is tolerated well (600mg oral daily D1, D2 & 25mg oral daily D3-D7), pulse dose escalation can continue as described above, with erlotinib at the daily low dose of 25 mg oral on D3-D7.
  Other Names: The assigned dosing schedule will be repeated weekly x 3 to complete a 3 week; (21 day) cycle. Cycle 1 will be 4 weeks to account for one week of lead in; pulse dose erlotinib only.

SUMMARY:
The purpose of this study is to test the safety of different ways of taking erlotinib. The investigators want to find out what effects, good and/or bad, combination daily low dose and twice weekly high dose erlotinib has on the patient and lung cancer. The investigators are also seeing whether different schedules of erlotinib are better at treating lung cancer that has spread to the central nervous system.

CNS expansion phase:

The pulse continuous regimen will be then assess in patients with EGFR mutant lung cancers and CNS involvement. An additional expansion cohort (A) will enroll 19 patients with newly diagnosed EGFR mutant lung cancer with CNS involvement at diagnosis. The patients in the expansion cohorts will undergo the same treatment plan as the patients in the dose expansion cohort. A patient in the expansion cohorts will not be replaced if he/she does not finish the first 28 day (cycle 1) treatment period.

ELIGIBILITY:
Inclusion Criteria:

* MSKCC pathologically-proven diagnosis locally advanced Stage III not amenable to definitive, curative treatment or Stage IV or recurrent non-small cell lung cancer
* Documented presence of EGFR mutation confirmed by MSKCC or a local facility.
* No prior treatment with erlotinib, gefitinib, or other EGFR tyrosine kinase inhibitors
* Age ≥ 18 years
* Measurable (RECIST 1.1) indicator lesion not previously irradiated.
* Karnofsky Performance Status ≥ 70%
* Ability to take oral medications
* A negative serum pregnancy test obtained within 4 weeks prior to the start of treatment in all women of child-bearing potential.
* All women of child bearing potential and sexually active men must agree to use adequate methods of birth control throughout the study which includes use of oral contraceptives with an additional barrier methods, double barrier methods, Depo-Provera, permanent sterilization of patient or partner or total abstinence.

Expansion A:

* brain metastases or leptomeningeal not previously treated with radiation or surgery

Exclusion Criteria:

* Inadequate recovery from any toxicity related to prior treatment (to Grade 2 or baseline).
* Inadequate hematologic function defined as ANC < 1000 cells/mm³, Platelet count <75,000/mm³ or Hemoglobin <9.0g/dL.
* Inadequate hepatic function defined by AST/ALT >3x upper limit of normal (ULN), Total bilirubin>2x ULN, Alkaline phosphatase >3x ULN.
* Symptomatic brain metastasis requiring radiation therapy or escalating doses of steroids.
* Patients with clinically stable brain metastases or leptomeningeal disease (previously treated or untreated) are eligible. Patients in expansion cohort A must have at least one untreated CNS lesion
* Women who are breastfeeding or pregnant.
* Any evidence of clinically active interstitial lung disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2013-10-15 (Actual); Primary Completion 2018-11-08 (Actual); Study Completion 2018-11-08 (Actual)

PRIMARY OUTCOMES:
to determine the maximum tolerated dose (MTD) | 1 year
  The study will use a standard 3+3 dose escalation design. Three to six patients will need to be enrolled at each dose level and assessed for DLT for 1 full cycle (28 days for cycle 1) before dose escalation decision is made.

SECONDARY OUTCOMES:
to evaluate the safety profile | 1 year
  Toxicity will be graded according to NCI CTCAE, version 4.0. The analysis of safety/tolerability data will be descriptive; toxicity events will be individually tabulated.
Progression Free Survival (PFS) | 1 year
  Progression free survival (PFS) is defined as the duration of time from first treatment to time of progression or death, whichever occurs first.
Response rate (RR) | 1 year
  sum of complete responses and partial responses according to RECIST 1.1
Overall survival (OS) | 1 year
  Overall survival (OS) is defined as the duration of time from first treatment to time of death.

CONTACTS AND LOCATIONS:
Overall Officials: Helena Yu, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Memoral Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Rockville Centre, Rockville Centre, New York
  - Memoral Sloan Kettering Cancer Center at Phelps, Sleepy Hollow, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/